CLINICAL TRIAL: NCT05529407
Title: Trial of Simple Vaginal Tampons vs Glass Vaginal Dilators in Treatment of Genitopelvic Penetration Disorder
Brief Title: Trial of SVTampons vs Glass Vaginal Dilators in Treatment of Vaginismus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe Filiz Gökmen Karasu, Doctor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bezmialem.5.22. 553
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-05

CONDITIONS: Vaginismus
Keywords: genitopelvic pain disorder, vaginismus
MeSH Terms: conditions — Vaginismus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Vaginal Tampon (Experimental): Dilation exercises will be performed with tampon
  Interventions: Device: Simple Vaginal Tampon
- Glass Vaginal Dilator (Experimental): Dilation exercises will be performed with vaginal dilator
  Interventions: Device: Glass Vaginal Trainer

INTERVENTIONS:
Device: Simple Vaginal Tampon — Use of single use vaginal tampons
  Other Names: SVT
  Arms: Simple Vaginal Tampon
Device: Glass Vaginal Trainer — Use of glass vaginal trainers
  Other Names: GVT
  Arms: Glass Vaginal Dilator

SUMMARY:
The aim of this study is to compare the success rates of vaginismus therapy using a tampon or a dilator during exposure

DETAILED DESCRIPTION:
Tampon Group

Exercises will be performed with tampon

Dilator Group

Exercises wil be performed with dilator

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant/non lactating women aged between 18-50
* diagnosed with primary vaginismus of Lamont level II or higher

Exclusion Criteria:

* hymenal abnormalities, congenital vaginal abnormalities, vulvodynia, secondary vaginismus following physical or psychological trauma, infection, menopausal period or pelvic pathology and with any psychiatric or physiological disease.
* Patients with husbands possessing a history of sexual dysfunction (erectile dysfunction or premature ejaculation, for example)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Sucessfull Intercourse-Diary | 30 days
  3 point scale: 1-did not try. 2- try but unseccesfull. 3- successfull intercourse

SECONDARY OUTCOMES:
GRISS: Golombuk Rust Inventory of Sexual Satisfaction | 30 day
  Higher scores indicate greater problems
FSFI Score | 30 day
  Higher scores indicate less problem
Fear of Coitus Subscale | 30 day
  Fear of sexuality

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslan M, Yavuzkir S, Baykara S. Is "Dilator Use" More Effective Than "Finger Use" in Exposure Therapy in Vaginismus Treatment? J Sex Marital Ther. 2020;46(4):354-360. doi: 10.1080/0092623X.2020.1716907. Epub 2020 Feb 13. PMID 32052704